CLINICAL TRIAL: NCT05355103
Title: Effects of an Educational Tool on Knowledge and Risk Retention About Epidural Analgesia in Parturients: a Prospective Before-and-after Study
Brief Title: Effects of an Educational Tool on Knowledge and Risk Retention About Epidural Analgesia in Parturients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie-Chantal Dubois, Clinical professor of anesthesiology, Université de Sherbrooke
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021-3575: Epid_Consent
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Analgesia, Epidural
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Women having received epidural analgesia after a standard verbal consent provided by the anesthesiologist before doing the epidural technique, representing the standard of practice in our institution
- Exposed group (Active Comparator): Woman having received epidural analgesia after having received and read an educational tool at her admission to labour and delivery unit, in addition to the standard verbal consent.
  Interventions: Other: Educational tool about epidural analgesia

INTERVENTIONS:
Other: Educational tool about epidural analgesia — See arm description
  Arms: Exposed group

SUMMARY:
The purpose of this study if to assess the basic knowledge of parturients about epidural analgesia, including an assessment of risks and benefits, but also risks associated with the procedure, and the impact of giving an informative document, in addition to usual consent counseling, on retention of risks.

A questionnaire was build by Delphi method by an expert panel in anesthesia. The questionnaire was answered on the first postpartum day by a group of patient that received the usual consent in the investigators's institution, including a standard explanation of risks and benefits at the moment they receive the epidural analgesia.

Parallel to the recruiting of the first group of patient receiving standard information and consent, an educational tool was build to provide informations relative to the epidural, including informations about the technique, the functioning of the epidural, the risks and benefits.

A second group of patient, who will received the educational tool antepartum at the time of admission to hospital for their delivery, will answer the same questionnaire on post-partum day 1. The results will then be compared to determine if the educational tool can improve the knowledge about epidural and so lead to a better consent about the epidural technique.

Comments about the educational tool and suggestions for improvement will also be collected.

DETAILED DESCRIPTION:
Discussing the risk and benefits of an epidural to a laboring woman can be a difficult task. Obtaining consent for the procedure whilst the pain, the anxiety, and the necessity of acting fast because of an active labor are added to the overwhelming quantity of information a laboring woman receive is among the challenges anesthesiologist must face before doing an epidural. The validity of the consent of a labouring women has already been proven in several studies. Indeed, it has been shown by that pain, either mild or severe, has no impact on the retention of epidural risks that have been explained. However, there is a significant variability regarding risk disclosure within different practice settings, particularly with respect to the incidence of serious complications. In studies, knowledge about the epidural and retention of information given at the time of consent remains poor, but could be improved by a learning tool (e.g., video, explanatory leaflet)

At the investigators's institution, standardized risks are exposed to the patient during the epidural technique. The five risks mentioned are hypotension, lumbar pain, failure (10%), risk of dura mater puncture (1%) and post-puncture headache as well as severe nerve injury up to paralysis (1/200 000). These risks are checked off on the anesthesia sheet when discussed with the patient. Groupe "before" will be asked about recall of risk and information giving after standard consent counseling. Groupe "after" will be exposed to an informative document explaining the risk as soon as active labour was confirmed. Participants will also have usual consent information standardized by local practice.

On post-partum day 1, participants will be asked about the risks exposed at the moment of consent regarding epidural analgesia by means of a questionnaire. The questionnaire distributed to patients contains true and false statement about the epidural and they will be asked about the truth of information. No additional information about the epidural will be disclose to the patients during the questionnaire. Group "before" will also be asked questions about how they would like to receive information concerning epidural and group "after" will be asked about if they appreciate receiving an informative brochure.

The informative document will be created by the study team and sent to the anesthesia and obstetrics teams in at study team's hospital for pre-approval. The maternity nurses will be asked to give the document as soon as the patient will be admitted to the ward. Before being recruited, parturient will have to ensure that they had indeed read the document before receiving epidural analgesia.

The aim of this before-and-after study is to evaluate the impact of adding an information document available at the admission for active labour on improving the knowledge of patients receiving epidural anesthesia as well as its effectiveness on retention of the risks explained at the time of consent. In addition, one of the sub-objectives is to identify which factors influence risk retention in order to eventually better adapt our pre-epidural counseling.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Age over 18 years old
* Had epidural analgesia during labour

Exclusion Criteria:

* Medical condition having influence on the risks of receiving epidural analgesia
* Insufficient understanding of french language
* Inability to provide medical consent
* Diagnosed and documented intellectual limitation
* Epidural anesthesia being converted to general anesthesia for a urgent cesarean section
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Knowledge and risk retention about epidural analgesia | Post-partum day 1
  Assessment of knowledge and risk retention about epidural analgesia. A questionnaire was build using Delphi method by an expert panel composed of anesthesiologists and Obstetric anesthesiologists. The final score of this questionnaire is the measurement tool for the primary outcome and is a dependant variable.
  * Score will be determined by the number of right answers a patient has on a scale of 0 to 12 (12 questions)
  * A patient gets 1 point for every right answer
  * The scale is based on the number of questions in the questionnaire and is not validated in the literature
  Since the two groups are independent, a T-test will be used if the data are normal. If not, a Mann-Whitney test will be used.
  Multivariates analysis by linear regression will be done for the variables above to consider possible confounding factors:
  * Previous epidural analgesia
  * Pain at the moment of the epidural technique
  * Satisfaction about the information received about epidural analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada